CLINICAL TRIAL: NCT01488071
Title: A Randomised, Double-blind, Parallel-group, Active-controlled, Flexible Dose Study Evaluating the Effects of [Vortioxetine] Lu AA21004 Versus Agomelatine in Adult Patients Suffering From Major Depressive Disorder With Inadequate Response to Antidepressant Treatment
Brief Title: A Study of Vortioxetine (Lu AA21004) in Comparison to Agomelatine in Adults Suffering From Major Depression With Inadequate Response to Previous Medication
Acronym: REVIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14178A; 2011-002362-21 (EudraCT Number)
Record Dates: First submitted 2011-11-29; First posted 2011-12-08 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Multimodal antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine; agomelatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine 10 mg or 20 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Agomelatine 25 mg or 50 mg (Active Comparator)
  Interventions: Drug: Agomelatine

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets, daily, orally
  Other Names: Brintellix®
  Arms: Vortioxetine 10 mg or 20 mg
Drug: Agomelatine — encapsulated tablets, daily, orally
  Other Names: Valdoxan®
  Arms: Agomelatine 25 mg or 50 mg

SUMMARY:
The objective of the present study is to evaluate whether vortioxetine (10 or 20 mg/day) is at least as effective as agomelatine (25 to 50 mg/day) in patients with depressive symptoms that showed inadequate response to Serotonin Reuptake Inhibitors (SRI) antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* The patient is being treated with a serotonin reuptake inhibitor (SRI) antidepressant (monotherapy) that was prescribed to treat Major Depressive Episode (DSM-IV-TR criteria)
* The response to the current SRI treatment is inadequate and patient agrees to discontinue the current SRI at the baseline
* Montgomery Åsberg Depression Rating Scale (MADRS) total score ≥22 at the Screening Visit and Baseline
* The patient, if a woman, must: agree not to try to become pregnant during the study, AND use adequate, highly effective contraception

Exclusion Criteria:

* The patient has any current Axis I disorders (DSM-IV criteria) other than Major Depressive Disorder (MDD), General Anxiety Disorder (GAD) and Social Anxiety Disorder (SAD)
* The patient is at significant risk of suicide
* The patient is currently receiving formal psychotherapy or other psychoactive medications

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Adair M, Christensen MC, Florea I, Loft H, Fagiolini A. Vortioxetine in patients with major depressive disorder and high levels of anxiety symptoms: An updated analysis of efficacy and tolerability. J Affect Disord. 2023 May 1;328:345-354. doi: 10.1016/j.jad.2023.01.074. Epub 2023 Jan 26. PMID 36708956
- [Derived] Papakostas GI, Nielsen RZ, Dragheim M, Tonnoir B. Efficacy and tolerability of vortioxetine versus agomelatine, categorized by previous treatment, in patients with major depressive disorder switched after an inadequate response. J Psychiatr Res. 2018 Jun;101:72-79. doi: 10.1016/j.jpsychires.2018.02.017. Epub 2018 Feb 22. PMID 29554497
- [Derived] Montgomery SA, Nielsen RZ, Poulsen LH, Haggstrom L. A randomised, double-blind study in adults with major depressive disorder with an inadequate response to a single course of selective serotonin reuptake inhibitor or serotonin-noradrenaline reuptake inhibitor treatment switched to vortioxetine or agomelatine. Hum Psychopharmacol. 2014 Sep;29(5):470-82. doi: 10.1002/hup.2424. PMID 25087600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In- or outpatients who had been treated with antidepressant selective serotonin reuptake inhibitor (SSRI) or selective noradrenaline reuptake inhibitor (SNRI) monotherapy that was prescribed to treat a single episode of Major Depressive Disorder (MDD) or recurrent MDD.
Pre-assignment Details: The study will consist of a screening period of 4 to 10 days before the Baseline Visit, followed by a 12-week treatment period with vortioxetine or agomelatine. A safety follow-up will be done approximately 4 weeks after the Completion/Withdrawal Visit.
Groups:
- Vortioxetine 10 mg or 20 mg; Agomelatine 25 mg or 50 mg: encapsulated tablets, daily, orally
Period: Overall Study
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Started | 253 (all-patients-treated set (APTS)) | 242 (APTS)
Completed | 200 | 179
Not Completed | 53 | 63
Not completed — Adverse Event | 15 | 23
Not completed — Lack of Efficacy | 11 | 17
Not completed — Non-compliance with study drug | 2 | 0
Not completed — Protocol Violation | 5 | 7
Not completed — Withdrawal of Consent | 14 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative or Other Reason(s) | 5 | 4

BASELINE CHARACTERISTICS:
Population: Age and Gender: All-patients-treated set (APTS) - all patients in the APRS who took at least one dose of investigational medicinal product (IMP).
  Study Specific Characteristics: Full-analysis set (FAS) - all patients in the APTS who had a valid baseline assessment and at least one valid post-baseline assessment of the MADRS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg | Total
Number analyzed (Participants) | 253 | 242 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.4) | 45.6 (12.4) | 46.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 175 | 370
  Male | 58 | 67 | 125
MADRS: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 - 60. The higher the score, the more severe.
  units on a scale | 29.1 (4.4) | 28.7 (4.0) | 28.9 (4.2)
HAM-A: Baseline Total Score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56; higher score indicates greater anxiety.
  units on a scale | 21.6 (6.3) | 21.4 (6.2) | 21.5 (6.2)
CGI-S Baseline Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating. Higher score indicates that the patient is more ill.
  units on a scale | 4.4 (0.6) | 4.4 (0.6) | 4.4 (0.6)
SDS Total Baseline Score [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
  units on a scale | 19.2 (5.3) | 19.3 (5.2) | 19.3 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score at Week 8
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 220 | 190
units on a scale | -16.53 (0.48) | -14.38 (0.51)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Non-Inferiority or Equivalence — Mixed model for repeated measurements (MMRM), using all available data, with a freely varying mean and covariance structures and with treatment, week, and site group as fixed factors and the baseline score as a covariate. The model also included interaction between week and baseline score, as well as interaction between week and treatment. Non-inferiority, upper limit of Confidence Interval should not exceed 2; p = 0.0018, Mixed Models Analysis — Under established non-inferiority the p-value is not adjusted; MMRM; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-3.51 to -0.81], Standard Error of Mean 0.69

2. Secondary Outcome: Change From Baseline in MADRS Total Score at Week 12
Time Frame: Baseline and Week 12
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 200 | 178
units on a scale | -18.95 (0.50) | -16.92 (0.53)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0054, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-3.45 to -0.60], Standard Error of Mean 0.72

3. Secondary Outcome: Change From Baseline in HAM-A Total Score at Week 8
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56; higher score indicates greater anxiety, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 220 | 190
units on a scale | -11.68 (0.39) | -9.79 (0.42)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-2.98 to -0.80], Standard Error of Mean 0.56

4. Secondary Outcome: Change From Baseline in HAM-A Total Score at Week 12
Time Frame: Baseline and Week 12
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 200 | 178
units on a scale | -13.52 (0.40) | -11.59 (0.42)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-3.04 to -0.81], Standard Error of Mean 0.57

5. Secondary Outcome: Change From Baseline in CGI-S Score at Week 8
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating. Higher score indicates that the subject is more ill, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 220 | 190
units on a scale | -1.84 (0.07) | -1.55 (0.07)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.48 to -0.11], Standard Error of Mean 0.10

6. Secondary Outcome: Change From Baseline in CGI-S Score at Week 12
Time Frame: Baseline and Week 12
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 200 | 178
units on a scale | -2.20 (0.07) | -1.93 (0.07)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0075, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.47 to -0.07], Standard Error of Mean 0.10

7. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment. Higher score = more affected.
Time Frame: Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 220 | 190
units on a scale | 1.97 (0.06) | 2.22 (0.07)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.08], Standard Error of Mean 0.09

8. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 12
Time Frame: Week 12
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 200 | 178
units on a scale | 1.74 (0.06) | 1.99 (0.07)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.07], Standard Error of Mean 0.09

9. Secondary Outcome: Proportion of Patients Who Respond at Week 8 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Baseline and Week 8
Population: FAS, last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 252 | 241
percentage of participants | 61.5 | 47.3
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0012, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.26 to 2.60]

10. Secondary Outcome: Proportion of Patients Who Respond at Week 12 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Baseline and Week 12
Population: FAS, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 252 | 241
percentage of participants | 69.8 | 56.0
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0014, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.26 to 2.65]

11. Secondary Outcome: Proportion of Patients Who Are in Remission at Week 8 (Remission is Defined as a MADRS Total Score <=10)
Time Frame: Week 8
Population: FAS, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 252 | 241
percentage of participants | 40.5 | 29.5
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0054, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.17 to 2.52]

12. Secondary Outcome: Proportion of Patients Who Are in Remission at Week 12 (Remission is Defined as a MADRS Total Score <=10)
Time Frame: Week 12
Population: FAS, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 252 | 241
percentage of participants | 55.2 | 39.4
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0002, Regression, Logistic — Wald's Test. No adjustments for multiple comparisons were made; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.39 to 2.90]

13. Secondary Outcome: Change From Baseline in SDS Total Score at Week 8
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Baseline and Week 8
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 162 | 135
units on a scale | -9.28 (0.53) | -7.06 (0.55)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -2.22, 95% CI 2-sided [-3.63 to -0.81], Standard Error of Mean 0.72

14. Secondary Outcome: Change From Baseline in SDS Total Score at Week 12
Time Frame: Baseline and Week 12
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 10 mg or 20 mg | Agomelatine 25 mg or 50 mg
Number analyzed (Participants) | 148 | 132
units on a scale | -10.99 (0.55) | -9.24 (0.58)
Statistical Analysis 1: Comparison: Vortioxetine 10 mg or 20 mg vs Agomelatine 25 mg or 50 mg; Test type: Superiority or Other; p = 0.0209, Mixed Models Analysis — No adjustments for multiple comparisons were made; The same MMRM methodology as for the primary endpoint was used; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.23 to -0.27], Standard Error of Mean 0.75

ADVERSE EVENTS:
Arm/Group | Vortioxetine | Agomelatine
Serious Adverse Events (participants affected / at risk) | 3/253 | 4/242
Other Adverse Events (participants affected / at risk) | 82/253 | 77/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vortioxetine (N=253) | Agomelatine (N=242)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0/195 | 1/175
Social stay hospitalisation (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=253) | Agomelatine (N=242)
Nausea (Gastrointestinal disorders) | 41 | 22
Dizziness (Nervous system disorders) | 18 | 28
Headache (Nervous system disorders) | 26 | 32
Somnolence (Nervous system disorders) | 10 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published. Authors of the primary publication based on this study must fulfil the criteria defined by the International Committee of Medical Journal Editors (ICMJE). The primary publication must be published before any secondary publications are submitted for publication.